CLINICAL TRIAL: NCT01384318
Title: Accuracy of Using the CPAP Technique to Eliminate Air Leak and Prevent Excessive Endotracheal Tube Cuff Pressures
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chairman Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Other Study IDs: IRB11-00414
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Surgical Patients Intubated With Cuffed ETT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cuffed ETT: Patients intubated with cuffed endotracheal tubes.
  Interventions: Other: Manometer

INTERVENTIONS:
Other: Manometer — Measuring cuff pressure

SUMMARY:
In common clinical practice, one means of ensuring an acceptable cuff pressure in endotracheal tubes (ETT) is to hold continuous positive airway pressure (CPAP) of 20-25 cmH2O and inflate the cuff of the ETT until no gas leak is noted around the cuff. The purpose of this study is to validate this technique by checking the intracuff pressure using a manometer after the cuff is inflated using the CPAP technique.

ELIGIBILITY:
Inclusion Criteria:

* Having a cuffed ETT placed per treating anesthesiologist
* < 18 yrs of age.

Exclusion Criteria:

* None

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients intubated with cuffed ETTs.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Cuff pressure | Baseline
  cm H2O measured by manometer

CONTACTS AND LOCATIONS:
Overall Officials: Joseph D Tobias, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Eschertzhuber S, Salgo B, Schmitz A, Roth W, Frotzler A, Keller CH, Gerber AC, Weiss M. Cuffed endotracheal tubes in children reduce sevoflurane and medical gas consumption and related costs. Acta Anaesthesiol Scand. 2010 Aug;54(7):855-8. doi: 10.1111/j.1399-6576.2010.02261.x. Epub 2010 Jun 15. PMID 20560884
- [Background] Weiss M, Dullenkopf A, Fischer JE, Keller C, Gerber AC; European Paediatric Endotracheal Intubation Study Group. Prospective randomized controlled multi-centre trial of cuffed or uncuffed endotracheal tubes in small children. Br J Anaesth. 2009 Dec;103(6):867-73. doi: 10.1093/bja/aep290. Epub 2009 Nov 3. PMID 19887533
- [Background] Weiss M, Dullenkopf A. Cuffed tracheal tubes in children: past, present and future. Expert Rev Med Devices. 2007 Jan;4(1):73-82. doi: 10.1586/17434440.4.1.73. PMID 17187473